CLINICAL TRIAL: NCT04022577
Title: Effects of Adherence Therapy on Medication Adherence in Patients With Schizophrenia Spectrum Disorder: A Randomized Controlled Trial
Brief Title: Effects of Adherence Therapy on Medication Adherence in Patients With Schizophrenia Spectrum Disorder
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Collaborators: Taipei Veterans General Hospital, Taiwan (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: YM108024E
Record Dates: First submitted 2019-07-10; First posted 2019-07-17 (Actual); Last update posted 2024-03-07 (Actual); Status verified 2023-10

CONDITIONS: Motivational Interviewing; Schizophrenia Spectrum Disorder; Medication Adherence
Keywords: Adherence Therapy; Insight; Medication Adherence; Motivational Interviewing; Schizophrenia Spectrum Disorder; Symptom severity; Randomized controlled trial
MeSH Terms: conditions — Medication Adherence | interventions — Motivational Interviewing; Control Groups

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): The experimental group will participate in a eight session course of Adherence Therapy
  Interventions: Behavioral: Adherence Therapy
- control group (Placebo Comparator): The control group received routine care
  Interventions: Behavioral: control group

INTERVENTIONS:
Behavioral: Adherence Therapy — Motivational interviewing-based AT in this study was based on Chien et al., (2016) and Gray et al., (2010) eight-session AT using the motivational interviewing technique (and principles of cognitive behavioral therapy).
  Other Names: Motivational interviewing
  Arms: experimental group
Behavioral: control group — The control group received routine care
  Arms: control group

SUMMARY:
This study will explore the effect of Adherence Therapy(AT) on medication adherence in patients with schizophrenia spectrum disorder.

DETAILED DESCRIPTION:
A single-blind, randomized controlled trial with a repeated-measures, two parallel groups design will be conducted for 120 participants with schizophrenia spectrum in regional hospital in northern Taiwan. After baseline data collection finished, the blocked randomization will be employed to assign participants to two groups. The experimental group will participate in a eight session course of Adherence Therapy. The control group received routine care. The data will be collected for baseline(T0) and after 4 session interim analysis(T1；9-12 weeks) and 8 session after intervention(T2；21-28 weeks). A structured Questionnaire will use to collect data on the Medication Adherence Rating Scale, Schedule for the Assessment of Insight, Internalized Stigma of Mental Illness Scale, Self-Appraisal of Illness Questionnaire and Positive and Negative Syndrome Scale. Data analysis will employ Statistical Package for the Social Sciences 20.0 with Generalized estimating equations approach to examine effects of Adherence Therapy and routine care on medication adherence.

ELIGIBILITY:
Inclusion Criteria:

* aged 20-64
* were Chinese speaking or Taiwanese speaking;
* diagnosed with schizophrenia or schizoaffective disorder
* recent history of non-adherence to antipsychotic medication.

  1. Non-adherence to medication was defined as a recent history of cessation of psychiatric admission for more than one month at a time
  2. The patient recently (half year) relapse of mental illness
  3. Family and Health care worker state that the patient has taken irregular medication
* demonstrated cognitive understanding of the research plan and provided consent.

Exclusion Criteria:

* discharged from hospital for at least 3 months
* no intellectual disability, organic brain diseases or Cognitive impairment
* no alcohol or sub-stance abuse problems
* were not attending medication management program .

Ages: 20 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Actual)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-08-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Medication Adherence Rating Scale | for two study groups at baseline(T0) and after 4 session interim analysis (T1；9-12 weeks) and 8 session after intervention (T2；21-28 weeks).
  The Medication Adherence Rating Scale was developed by Thompson et al. (2000). It evaluates the adherence behavior and attitude of the patient within the previous week. There are 10 close-ended questions (yes/no answers) in the questionnaire.

SECONDARY OUTCOMES:
Schedule for the Assessment of Insight, SAI | for two study groups at baseline(T0) and after 4 session interim analysis(T1；9-12 weeks) and 8 session after intervention(T2；21-28 weeks).
  The Schedule of Assessment of Insight (SAI) measures multiple dimensions of insight, including compliance with treatment, recognition of illness, re-labeling of psychotic phenomena, and awareness of changes in mental functioning and psychosocial consequences of the illness.The maximum score of the SAI is 14, with higher SAI scores indicating greater insight. The Cronbach alpha for the SAI was 0.96, and inter-rater reliability (r) between the two research psychiatrists was .92 in the present study.
Positive and Negative Syndrome Scale, PANSS | for two study groups at baseline(T0) and after 4 session interim analysis(T1；9-12 weeks) and 8 session after intervention(T2；21-28 weeks).
  PANSS assessed the severity of psychotic symptoms in terms of three subscales, including positive symptoms (hallucinations,delusional beliefs, and 30-item 7point Likert scale (from 1-'Absent' to 7-'Extremely').
Self-Appraisal of Illness Questionnaire, SAIQ | for two study groups at baseline(T0) and after 4 session interim analysis(T1；9-12 weeks) and 8 session after intervention(T2；21-28 weeks).
  The Self-Appraisal of Illness Questionnaire (SAIQ) was used to assess patients' insight into their illness.The need for treatment and presence/outcome of illness subscales of SAIQ have been used as brief screening instruments for schizophrenic patients who may be at risk for treatment noncompliance. Lower SAIQ subscale scores indicate reduced awareness of the psychiatric illness. This scale is a self reporting instrument composed of 17 items in which participants are asked to rate the extent to which they agreed with each statement by using a 4-point Likert scale ranging from 0 (ie, "do not agree at all") to 3 (ie, "agree completely").
  The internal consistency of the scale was 0.867, and the retest reliability was 0.82.

CONTACTS AND LOCATIONS:
Overall Officials: Yan Laing Chen, BSN, Study Chair — Institute of Community Health Care National Yang-Ming University
Locations (1):
- National Yang-Ming University, Taipei, Taiwan